CLINICAL TRIAL: NCT05828823
Title: Comparative Effectiveness of an Individualized Model of Hemodialysis Versus Conventional Hemodialysis
Brief Title: Incremental Hemodialysis: The TwoPlus Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00092986; CER-2022C1-26300 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-03-29; First posted 2023-04-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: End-Stage Kidney Disease
Keywords: Hemodialysis; Clinically-Matched Incremental Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a randomized parallel-group type 1 hybrid study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clinically-matched Incremental Hemodialysis ( CMIHD) (Experimental): Randomized group to have hemodialysis prescription tailored based on residual kidney function and clinical manifestations starting at twice weekly.
  Interventions: Device: Hemodialysis twice weekly
- Conventional Hemodialysis (CHD) (Active Comparator): Randomized group to conventional three times a week hemodialysis.
  Interventions: Other: Hemodialysis thrice weekly

INTERVENTIONS:
Device: Hemodialysis twice weekly — Frequency and duration of hemodialysis is tailored to the patient. Adjuvant pharmacotherapy is prescribed to maintain volume, electrolyte and acid-base homeostasis ( e.g., diuretics, sodium bicarbonate and potassium binding patiromer)
  Arms: Clinically-matched Incremental Hemodialysis ( CMIHD)
Other: Hemodialysis thrice weekly — Conventional hemodialysis regimen
  Arms: Conventional Hemodialysis (CHD)

SUMMARY:
This study is to prospectively compare clinical effectiveness between clinically- matched incremental hemodialysis and conventional hemodialysis in patients with incident kidney dysfunction requiring dialysis and residual kidney function.

The study will enroll 350 patients on chronic hemodialysis and 140 caregivers of enrolled patients. Patients will be randomized in 1:1 ratio to either incremental start hemodialysis or conventional hemodialysis. Caregivers will be followed along with patients for an average period of 2 years post randomization.

DETAILED DESCRIPTION:
This study will analyze the effects of differentiated care with individualized hemodialysis on patient health related quality of life, fatigue, employment, and caregiver burden in patients with Kidney dysfunction requiring dialysis (KDRD) and appreciable kidney function.

This study will compare the outcomes in survival, hospitalization, preservation of the kidney function and quality of life between hemodialysis tailored to each patient needs (incremental) and conventional hemodialysis.

ELIGIBILITY:
Patient eligibility Criteria:

Inclusion Criteria:

* Clinical Inclusion Criteria:
* Age ≥ 18 years
* Incident kidney dysfunction requiring dialysis (KDRD) started on maintenance, in-center hemodialysis (HD), or anticipated to be started on maintenance, in-center HD within the next 12 weeks
* Has received ≤36 sessions of intermittent HD (i.e., on HD for ≤12 weeks) at the time patient is approached for potential study participation

Residual Kidney Function Inclusion Criteria:

* Kidney urea clearance <2.0 mL/min
* Urine volume# of ≥500 mL/24 h

Exclusion Criteria:

* Pre-HD serum K ≥5.8 mEq/L, Na ≤125 mEq/L, or bicarbonate level ≤17 mEq/L
* Requirement or anticipated requirement of high-volume ultrafiltration
* Unable or unwilling to follow the study protocol for any reason
* Known pregnancy or planning to attempt to become pregnant or lactating women
* Estimated survival or dialysis modality change or center transfer <6 months

Caregiver Eligibility Criteria:

* be at least 18 years old
* be the main caregiver (at patient's choice)
* be a close relative of the patient (spouse, child, sibling, parent, grandchild)
* have no known psychiatric and neurologic disorders (through direct inquiry from the person)
* not be a member of the medical or healthcare team
* not be the caregiver for another patient with chronic illness
* not have experienced severe life events within prior 3 months of enrollment (through direct inquiry from the person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Clinical events of safety | year 2
  composite of all-cause Emergency Department visits, hospitalizations, or death

SECONDARY OUTCOMES:
EuroQOL-5D-5L scores Health-related quality of life Health-related quality of life and residual kidney function | year 2
  Compare the effects of CMIHD and CHD - The descriptive system covers 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems - Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead.
Trail Making Test B scores Health-related quality of life Health-related quality of life and residual kidney function | Baseline and months 6, 12, 18, & 24
  Patient participants' cognitive function will be assessed using change in Trail Making Test B score - The Trail Making Test measures your visual attention, mental flexibility, processing speed, and motor speed based on how quickly and accurately you connect dots in ascending order (either numerically or with alternating numbers and letters). The test can be used to diagnose dementia and other cognitive disorders - Higher scores indicate a higher degree of cognitive impairment
Standardized Outcomes in Nephrology (SONG) scores Health-related quality of life Health-related quality of life and residual kidney function | Baseline and months 6, 12, 18, & 24
  SONG-HD Fatigue score - The SONG-HD Fatigue measure consists of three items that assess (1) the effect of fatigue on life participation, (2) tiredness, and (3) level of energy. These dimensions are assessed on a four-point Likert scale indicating increasing severity, ranging from zero (not at all) to three (severely). Higher scores meaning higher severity
Time to recover from hemodialysis (HD) Health-related quality of life Health-related quality of life and residual kidney function | Baseline and monthly up to 2 years
  Patient-reported functional status and fatigue will be assessed using Time to recover from HD
Caregiver burden Zarit Caregiver Burden Scores Health-related quality of life Health-related quality of life and residual kidney function | Baseline, months 6, 12, 18, & 24
  Caregiver burden will be assessed using the Zarit Caregiver Burden Scale - The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. 9. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Change in urine output | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, and Year 2
  Urine collections will be analyzed at the lab used by the dialysis center
Change in kidney urea clearance (mL/min/1.73 m2) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, and Year 2
  Urine collections will be analyzed at the lab used by the dialysis center
Change in kidney creatinine clearance (mL/min/1.73 m2) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, and Year 2
  Urine collections will be analyzed at the lab used by the dialysis center
Hospital free days per 100 patient-days | year 2
  The duration of hospital-free days will be determined for each patient and calculated in the whole cohort per 100 patient-days. It is anticipated an array of hospitalization events for each participant, ranging from no hospitalization to frequent hospitalizations per study period. All periods of hospitalization, per each participant, will be analyzed. A period of hospitalization will be computed from date of hospital admission to the date of discharge. Hospital-free days may include one or more discrete time segments of non-hospitalization between periods hospitalization. The total hospital-free days per patient participant will be calculated as total study days - hospitalization days. Hospital-free days will be normalized per 100 patient-days.
Illness Intrusiveness Rating Scale | Assessed at baseline and monthly up to 2 years
  Patients will rate the degree of interference caused by HD treatments on the following domains: health, diet, work, active and passive recreation, financial situation, relationship with spouse, sex life, family and other social relations, self-expression/self- improvement, religious expression, and community/civic involvement. Individual item ratings and the sum across ratings will be recorded. The total scale has a range of 13 (minimum intrusiveness) to 91 (extreme intrusiveness).
Employment status | Baseline and months 6, 12, 18 and 24
  The employment status for patients and caregivers will be assessed through surveys.

OTHER OUTCOMES:
Characterize implementation processes using mixed methods - Intervention characteristics | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - External factors that mediate implementation | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - Adoption | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - Reach | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention
Characterize implementation processes using mixed methods - Sustainability, to assess barriers and facilitators to maintaining intervention | 2 years
  Process evaluation will include a) Intervention characteristics, to assess organizational readiness to change, intervention acceptability and appropriateness; b) Inner setting characteristics, to assess barriers and facilitators to the adoption of HD intervention at the partnering organizations; c) External factors that mediate implementation; d) Adoption; e) Reach; f) Fidelity, to assess adherence to serial timed urine collection and HD treatment schedule; and g) Sustainability, to assess barriers and facilitators to maintaining intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Murea, MD, Principal Investigator — Wake Forest Health Sciences; Peter Kotanko, Principal Investigator — Renal Research Institute
Locations (10):
- United States (10):
  - University of Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University School of Medicine (JHUSM), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Renal Research Institute (RRI), New York, New York
  - Northwell Health, Queens, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Virginia (UVA), Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Available upon investigator request

REFERENCES:
- [Derived] Murea M, Foley KL, Gautam SC, Flythe JE, Raimann JG, Abdel-Rahman E, Awad AS, Niyyar VD, Kovach C, Roberts GV, Jefferson NM, Conway PT, Rosales LM, Woldemichael J, Sheikh HI, Raman G, Huml AM, Knicely DH, Hasan I, Makadia B, Lea J, Daugirdas JT, Gencerliler N, Divers J, Kotanko P; TwoPlus Research Consortium; Nwaozuru UC. Protocol for the process evaluation of a randomised clinical trial of incremental-start versus conventional haemodialysis: the TwoPlus study. BMJ Open. 2025 Nov 28;15(11):e094392. doi: 10.1136/bmjopen-2024-094392. PMID 41314824
- [Derived] Murea M, Raimann JG, Divers J, Maute H, Kovach C, Abdel-Rahman EM, Awad AS, Flythe JE, Gautam SC, Niyyar VD, Roberts GV, Jefferson NM, Shahidul I, Nwaozuru U, Foley KL, Trembath EJ, Rosales ML, Fletcher AJ, Hiba SI, Huml A, Knicely DH, Hasan I, Makadia B, Gaurav R, Lea J, Conway PT, Daugirdas JT, Kotanko P; Two Plus Research Consortium. Comparative effectiveness of an individualized model of hemodialysis vs conventional hemodialysis: a study protocol for a multicenter randomized controlled trial (the TwoPlus trial). Trials. 2024 Jun 28;25(1):424. doi: 10.1186/s13063-024-08281-9. PMID 38943204